CLINICAL TRIAL: NCT03064321
Title: Self-Management, Insomnia, and Glucose Control in Adults With Diabetes
Brief Title: Diabetes Sleep Treatment Trial for Insomnia
Acronym: DSTT-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Eileen R. Chasens, Associate Professor of Nursing, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K24NR016685-01A1 (NIH)
Record Dates: First submitted 2017-02-15; First posted 2017-02-27 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Insomnia; Diabetes Mellitus, Type 2
Keywords: cognitive behavioral treatment
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Two group design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insomnia Intervention (Experimental): Insomnia intervention delivered via web using Cognitive Behavior Treatment
  Interventions: Behavioral: Insomnia Intervention
- Information Control (Other): General health information website
  Interventions: Other: Information Control

INTERVENTIONS:
Behavioral: Insomnia Intervention — The SHUTi intervention is based on a cognitive behavioral treatment for insomnia (CBT-I) and organized into six structured, weekly online sessions. Each week the participants will complete a 30-minute interactive learning module and to complete daily online sleep diaries will be used.
  Arms: Insomnia Intervention
Other: Information Control — Information on websites that are general health promoting
  Arms: Information Control

SUMMARY:
This study will test the effect of the an insomnia intervention with cognitive behavioral treatment delivered via web compared with an information control group on glucose control and self management behavioral in a sample of persons with type 2 diabetes (T2DM).

DETAILED DESCRIPTION:
Recent evidence supports that insomnia is a prevalent problem among persons with type 2 diabetes that may be associated with increased daytime sleepiness and fatigue, increased diabetes-related distress, decreased self-management behavior, and worse glycemic control. The main hypothesis of the current application is that a web-based cognitive behavioral treatment of insomnia (Sleep Health Using the Internet: SHUTi) in persons with T2DM will not only improve their nighttime sleep, but also improve their ability to integrate diabetes education into their daily behavior and positively affect their glucose control compared to a web-based Information Control (IC) group. The aims of this study are to 1) obtain preliminary data to facilitate further hypothesis development and enhance the feasibility of conducting a randomized clinical trial to examine if treatment of insomnia results in participant's being better able to integrate diabetes education into their self-management behavior and result in improved glucose control, 2) explore the associations among changes in insomnia severity, fatigue, daytime sleepiness, sleep quality, A1C (a measure of glucose control over the last three months) and diabetes self-management (DSM) behaviors, 3) explore average pre-intervention to post-intervention changes in insomnia severity, daytime symptoms (fatigue, sleepiness, mood) and DSM behaviors (diet and physical activity) in subjects treated with SHUTi + DSM compared to IC + DSM subjects at 3 months, and 4) explore sleep fragmentation as a potential physiological mechanism linking impaired glucose control (A1C) and sleep in subjects with insomnia and T2DM at baseline and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* (1) T2DM with suboptimal glucose control
* (2) age 18 years or older;
* (3) willing to be randomized to SHUTi or IC group;
* (4) able to speak, read, and write in English, and
* (5) insomnia symptoms with at least one daytime consequence [e.g. impaired mood, poor sleep quality, excessive daytime sleepiness, fatigue].

Exclusion Criteria:

* Type 1 or gestational diabetes
* Change in oral medications or > 10% change in insulin in last 3 months
* Acute medical or psychiatric illness or hospitalization ≤ 3 months (such as angina, stroke, major surgery, major depression or serious psychiatric conditions)
* AHI (apnea-hypopnea index; apnea [cessation of breathing] or hypopnea [reduction in breathing]) ≥ 10 episodes an hour on overnight sleep study
* Non-ambulatory
* Self-reported epilepsy, psychotic or bipolar disorder
* History of near-miss or auto accident during last 12 months
* Employed in safety sensitive job (e.g. truck driver or airline pilot)
* Working nights or rotating shifts
* Regular use of alerting (e.g., modafinil) medications
* Consumption of alcohol: Men: > 4 drinks a day or > 14 drinks per week
* Women: > 3 drinks a day or > 7 drinks per week
* If using sleep medications, the drug and/or dose changed in the past month
* Depression
* Medications for psychotic or bipolar disorders
* No internet access
* Pregnant or intend to become pregnant in the next four months (postmenopausal or confirmed not pregnant by a urine pregnancy test)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Average Glucose Control for Last 3 Months Assessed by A!C level | After 12 weeks of either the insomnia intervention or the information control intervention
  A1C level

SECONDARY OUTCOMES:
Sleep Quality | After 12 weeks of either the insomnia intervention or the information control intervention
  Scores on the Pittsburgh Sleep Quality Index questionnaire

OTHER OUTCOMES:
Insomnia Severity | After 12 weeks of either the insomnia intervention or the information control intervention
  Scores on the Insomnia Severity Index questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eileen R Chasens, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh School of Nursing, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No